CLINICAL TRIAL: NCT05415293
Title: Serum Docosahexaenoic Acid After Third Trimester Commercially Available Supplementation: a Randomized Clinical Trial
Brief Title: Commerical DHA Supplementation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI has confirmed there are no results because the samples were degraded.
Sponsor: University of New Mexico (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, Ellen Mozurkewich, Co-investigator, University of New Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mozurkewich 10-417; UL1RR031977 (NIH)
Record Dates: First submitted 2014-06-10; First posted 2022-06-13 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Randomized Clinical Trial; Docosahexaenoic Acid; Pregnancy
Keywords: docosahexaenoic acid; pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Expecta 200mg DHA supplement (Active Comparator): Women receive one daily softgel 200mg DHA algae-based DHA supplement sold as "Expecta."
  Interventions: Dietary Supplement: Expecta 200mg DHA
- Promise 275mg DHA supplement (Active Comparator): Women receive one daily softgel 275mg DHA fish oil-based DHA supplement sold as "Promise."
  Interventions: Dietary Supplement: Promise 275mg DHA
- Control/ no supplement (No Intervention): Women received care as usual and did not take any DHA supplement.

INTERVENTIONS:
Dietary Supplement: Expecta 200mg DHA
  Other Names: algae DHA
  Arms: Expecta 200mg DHA supplement
Dietary Supplement: Promise 275mg DHA
  Other Names: fish oil DHA
  Arms: Promise 275mg DHA supplement

SUMMARY:
The purpose of this study is to compare blood levels of women who take commericially available, low dose docosahexaenoic acid (DHA) dietary supplements in pregnancy with women who do not take supplements.

DETAILED DESCRIPTION:
The investigators recruited 73 pregnant women in the late third trimester from a low-risk midwifery clinic in compliance with the protocol approved by the investigators institutional review board regulations (HRPO #10-417). All women in the clinic were offered participation and enrollment was performed at 34-36 weeks gestational age for those who agreed. Exclusion criteria included, preeclampsia, gestational diabetes or pre-gestational diabetes, chronic use of medications, and other medical complication of pregnancy. Maternal data including age, gravidity, parity, gestational age, ethnicity, BMI at delivery, and mode of delivery were collected in compliance with the Health Insurance Portability and Accountability Act guidelines. Neonatal data, including gender, birth weight, height, and head circumference and maternal delivery charactersitics were collected after reviewing the delivery record.

Subjects consented to randomization into a group receiving a fish oil based 275mg Promise DHA (Biotegrity; Granbury, TX) by mouth each day, or an algae-based 200mg Expecta DHA (Mead Johnson; Evansville, IN) by mouth each day, or dietary habits as usual. Randomization assignments were concealed in opaque envelopes and revealed at the time of enrollment. Calendars were kept to document supplement use and unused supplements were turned in at the time of admission to labor and delivery. Pill counts were performed to verify the accuracy of calendars.

Sample size considerations: The investigators primary outcome measure was DHA level in maternal serum and neonatal cord blood. To detect a 15% increase in DHA proportions, it would require a sample size of 19 in each group. This study is a pilot investigation, designed to determine if a larger supplementation study would be feasible in the investigators population.

Collection of blood samples A venous blood sample was collected from each participant at the time of enrollment and randomization. Maternal blood was drawn from the antecubital fossa in tubes containing EDTA and stored at -4 degrees C. A second maternal sample was retrieved at the time of admission for labor in a similar fashion. Neonatal samples were similarly collected at the time of delivery, just after cord clamping. Within 72 hours of collection, nonhemolyzed maternal and neonatal samples were identified and centrifuged for 5 minutes in a clinical centrifuge, and the plasma portion was extracted and stored in 2-mL vials at -78 degrees C until fatty acid analysis was performed.

Fatty acid analyses:

Samples were allowed to thaw at room temperature and lipid extraction was performed using chloroform/methanol (2:1, v/v) according to the method of Folch et al (1957). The extracted lipid residue was weighed after drying at 45oC under a stream of nitrogen. The total phospholipid component of serum was isolated by silicic acid column chromatography (26) of the total lipid fraction obtained by extracting a 1-mL aliquot of serum with chloroform: methanol (2:1,v/v). Fatty acids were transesterified to generate methyl esters using 0.5 N NaOH in methanol and 14% (w/v) boron trifluoride in methanol (27). Undecenoic acid (Nu-Check Prep, Elysian, MN) was added prior to methylation, and served as an internal standard.

Fatty acid methyl esters were quantified using a gas chromatograph (6890N, Agilent Technologies, Sunnyvale, CA) equipped with an autoinjector, a split/splitless capillary injection system, and a flame ionization detector as described elsewhere(28)(). A customized fatty acid mixture described by Loor and Herbein (28) and made with pure methyl ester standards, including AA and DHA, (Nu-Check Prep, Elysian, MN, USA; Sigma, St. Louis, MO, USA) was used to identify peaks and determine response factors for integration with a Chem DataStation (Agilent Technologies, Sunnyvale, CA).

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant
2. 34-36 weeks gestational age

Exclusion Criteria:

1. Maternal medical disease
2. Gestational diabetes
3. Pre-eclampsia
4. Fetal anomalies
5. Ingestion of DHA or fish oil dietary supplements during the current pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Maternal serum DHA weight % at delivery | 5 months
  Weight proportion of DHA in the total plasma phospholipids after supplementation
DHA in newborn cord blood after supplementation | up to 72 hours
  Weight proportion of DHA in the total plasma phospholipids of newborn cord blood after maternal supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Steffen A Brown, MD, Study Director — University of New Mexico; Ellen L Mozurkewich, MD, MS, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico Hospital, Albuquerque, New Mexico, United States

REFERENCES:
- [Background] Wolfe MD, Chuang LT, Rayburn WF, Wen PC, VanderJagt DJ, Glew RH. Low fatty acid concentrations in neonatal cord serum correlate with maternal serum. J Matern Fetal Neonatal Med. 2012 Aug;25(8):1292-6. doi: 10.3109/14767058.2011.631064. Epub 2012 Apr 24. PMID 22023348